CLINICAL TRIAL: NCT03330288
Title: Prospective Multicenter Non-interventional Study in Patients With Knee or Hip Osteoarthritis Having a Theraflex® Treatment to Evaluate Changes in Pain, Functions in Daily Living, and Quality of Life for an Observation Period up to 64 Weeks
Brief Title: Prospective Multicenter Non-interventional Study in Patients With Knee or Hip Osteoarthritis Having a Theraflex Treatment
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19649
Record Dates: First submitted 2017-10-06; First posted 2017-11-06 (Actual); Results first posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with Stage I-III Knee osteoarthritis (KOA): Participants were receiving Theraflex not earlier than 2 weeks prior to enrollment
  Interventions: Drug: Theraflex, BAY 874017
- Participants with Stage I-III Hip osteoarthritis (HOA): Participants were receiving Theraflex not earlier than 2 weeks prior to enrollment
  Interventions: Drug: Theraflex, BAY 874017

INTERVENTIONS:
Drug: Theraflex, BAY 874017 — The first three weeks which do have a different posology (3 capsules a day) according to the label should be entered as a distinct period to the treatment period with a recommended posology of 2 capsules a day

SUMMARY:
The main purpose of this study is to evaluate how a long-term treatment with Theraflex during 64 weeks affects pain intensity in the affected knee or hip joint, the activity in daily living, the quality of life and patient satisfaction with treatment.

DETAILED DESCRIPTION:
Other information that is planned for evaluation in this study includes consumption of Theraflex, intake of analgesics for joint pain relief and description of basic patient characteristics such as age, weight and body mass index and others.

ELIGIBILITY:
Inclusion Criteria:

* Patients 45 to 75 years with Hip or Knee OA stage I to III
* Patient started current treatment with Theraflex not more than 2 weeks prior to inclusion into the study
* Personally signed and dated informed consent

Exclusion Criteria:

* Patients participating in an investigational program with interventions outside of routine clinical practice
* Patients with Hip or Knee OA stage 0 or stage IV
* Patients who have both Hip and Knee OA and OA of any other location
* Contraindications for use of Theraflex in accordance with approved label(known hypersensitivity, severe chronic renal failure)
* Females who are pregnant or breastfeeding
* Patients who completed a treatment with Theraflex or another combination of Gl+ Ch less than 5 months before start of the current treatment
* Patients who completed intra-articular corticosteroids treatment in the last 3 months to exclusion criteria
* Patients who completed hyaluronic injections of the lower limbs in the last 6 months

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who will be made aware about the study either by the treating physician OR by a pharmacist where a patient is purchasing Theraflex
Sampling Method: Non-Probability Sample
Enrollment: 1102 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-07-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Sci-Res Institute of Rheumatology n.a. V.A. Nasonova of RAMS, Moscow
  - Many locations, Multiple Locations

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 51 centers in Russian Federation, between 20-Nov-2017 (first participant first visit) and 13-Jul-2020 (Database clean). The Primary Completion date is 18-Mar-2020 (last participant last visit)
Pre-assignment Details: A total of 1111 participants were screened over the course of the study, of which 1102 participants were enrolled in the study. Among them, 824 participants were diagnosed with knee osteoarthritis (KOA), while 278 participants were diagnosed with hip osteoarthritis (HOA).
Period: Overall Study
Arm/Group | Participants With Stage I-III Knee Osteoarthritis (KOA) | Participants With Stage I-III Hip Osteoarthritis (HOA)
Started | 824 (Enrolled) | 278 (Enrolled)
Completed | 794 | 270
Not Completed | 30 | 8
Not completed — Other reason | 1 | 1
Not completed — Switching to a different disease-modifying delayed-release drug SYSADOA | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 26 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Stage I-III Knee Osteoarthritis (KOA) | Participants With Stage I-III Hip Osteoarthritis (HOA) | Total
Number analyzed (Participants) | 824 | 278 | 1102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (6.9) | 60.3 (7.21) | 60.4 (6.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 728 | 240 | 968
  Male | 96 | 38 | 134
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 820 | 278 | 1098
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Pain intensity subscale [Mean (Standard Deviation); unit: Scores on a scale] — KOA patients used KOOS questionnaire, HOA patients used HOOS questionnaire. Pain intensity is one subscale of KOOS and HOOS questionnaire, each pain intensity question provides standard answer options: 0=None, 1=Mild, 2=Moderate, 3=Severe, 4=Extreme. The results for KOOS pain intensity subscale were calculated as [100 - (mean value of all subscale questions * 100) / 4]. Results score is from 0 to 100. 100 indicating no symptoms and 0 indicating extreme symptoms. HOOS pain intensity subscale results calculation used a similar method. Population: KOA patients and HOA patients are reported separately for each Arm of the study
  Scores on a scale | 61.48 (16.434) | 60.97 (17.321) | NA (NA) — Two groups used different scales, so no output for total analysis.
Other symptom subscale [Mean (Standard Deviation); unit: Scores on a scale] — KOA patients used KOOS questionnaire, HOA patients used HOOS questionnaire. Other symptoms is one subscale of KOOS and HOOS questionnaire, each other symptoms question provides standard answer options: 0=None, 1=Mild, 2=Moderate, 3=Severe, 4=Extreme. The results for KOOS other symptoms subscale were calculated as [100 - (mean value of all subscale questions * 100) / 4]. Results score is from 0 to 100. 100 indicating no symptoms and 0 indicating extreme symptoms. HOOS other symptoms subscale results calculation used a similar method. Population: KOA patients and HOA patients are reported separately for each Arm of the study
  Scores on a scale | 62.25 (18.034) | 61.17 (17.691) | NA (NA) — Two groups used different scales, so no output for total analysis.
Functional activity of the joint subscale [Mean (Standard Deviation); unit: Scores on a scale] — KOA patients used KOOS questionnaire, HOA patients used HOOS questionnaire. Functional activity is one subscale of KOOS and HOOS questionnaire, each functional activity question provides standard answer options: 0=None, 1=Mild, 2=Moderate, 3=Severe, 4=Extreme. The results for KOOS functional activity subscale were calculated by converting value of all subscale questions to KOOS-Physical Short form score. Results score is from 0 to 100, 100 indicating no symptoms and 0 indicating extreme symptoms. HOOS functional activity subscale results used a similar method with HOOS-Physical Short form. Population: KOA patients and HOA patients are reported separately for each Arm of the study
  Scores on a scale | 61.46 (10.599) | 65.57 (16.515) | NA (NA) — Two groups used different scales, so no output for total analysis.
Life quality subscale [Mean (Standard Deviation); unit: Scores on a scale] — KOA patients used KOOS questionnaire, HOA patients used HOOS questionnaire. Life quality is one subscale of KOOS and HOOS questionnaire, each life quality question provides standard answer options: 0=None, 1=Mild, 2=Moderate, 3=Severe, 4=Extreme. The results for KOOS life quality subscale were calculated as [100 - (mean value of all subscale questions * 100) / 4]. Results score is from 0 to 100. 100 indicating no symptoms and 0 indicating extreme symptoms. HOOS life quality subscale results calculation used a similar method. Population: KOA patients and HOA patients are reported separately for each Arm of the study
  Scores on a scale | 44.99 (17.009) | 46.79 (17.507) | NA (NA) — Two groups used different scales, so no output for total analysis.
Patient satisfaction assessment [Mean (Standard Deviation); unit: Scores on a scale] — Patient satisfaction questionnaire was filled out during the visit to a doctor. A patient assessed treatment satisfaction against the Likert response scale : 5-very satisfied, 4-Satisfied, 3- No answer, 2-Dissatisfied, 1-very dissatisfied
  Scores on a scale | 3.2 (0.5) | 3.1 (0.42) | 3.1 (0.48)

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Pain Intensity Subscale
Description: KOA patients used KOOS questionnaire, HOA patients used HOOS questionnaire. Pain intensity is one subscale of KOOS and HOOS questionnaire, each pain intensity question provides standard answer options: 0=None, 1=Mild, 2=Moderate, 3=Severe, 4=Extreme. The results for KOOS pain intensity subscale were calculated as [100 - (mean value of all subscale questions * 100) / 4]. Results score is from 0 to 100. 100 indicating no symptoms and 0 indicating extreme symptoms. HOOS pain intensity subscale results calculation used a similar method.
Time Frame: From enrollment up to 64 weeks
Population: The outcome measure was analyzed based on participants who has KOOS/HOOS assessment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants With Stage I-III Knee Osteoarthritis (KOA) | Participants With Stage I-III Hip Osteoarthritis (HOA)
Number analyzed (Participants) | 824 | 278
Scores on a scale
  From Visit 1(enrollment) to Visit 2 (Week 16-24): number analyzed (Participants) | 798 | 272
  From Visit 1(enrollment) to Visit 2 (Week 16-24) | 18.07 (16.900) | 15.59 (16.686)
  From Visit 1(enrollment) toVisit 3 (Week 36-44): number analyzed (Participants) | 794 | 271
  From Visit 1(enrollment) toVisit 3 (Week 36-44) | 20.92 (17.946) | 20.06 (17.686)
  From Visit 1(enrollment) toVisit 4 (Week 56-64): number analyzed (Participants) | 794 | 270
  From Visit 1(enrollment) toVisit 4 (Week 56-64) | 22.87 (18.815) | 22.81 (19.550)

2. Primary Outcome: Changes in Other Symptoms Subscale
Description: KOA patients used KOOS questionnaire, HOA patients used HOOS questionnaire. Other symptoms is one subscale of KOOS and HOOS questionnaire, each other symptoms question provides standard answer options: 0=None, 1=Mild, 2=Moderate, 3=Severe, 4=Extreme. The results for KOOS other symptoms subscale were calculated as [100 - (mean value of all subscale questions * 100) / 4]. Results score is from 0 to 100. 100 indicating no symptoms and 0 indicating extreme symptoms. HOOS other symptoms subscale results calculation used a similar method.
Time Frame: From enrollment up to 64 weeks
Population: The outcome measure was analyzed based on participants who has KOOS/HOOS assessment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants With Stage I-III Knee Osteoarthritis (KOA) | Participants With Stage I-III Hip Osteoarthritis (HOA)
Number analyzed (Participants) | 824 | 278
Scores on a scale
  From Visit 1(enrollment) to Visit 2 (Week 16-24): number analyzed (Participants) | 798 | 272
  From Visit 1(enrollment) to Visit 2 (Week 16-24) | 15.48 (17.465) | 12.65 (16.937)
  From Visit 1(enrollment) toVisit 3 (Week 36-44): number analyzed (Participants) | 794 | 271
  From Visit 1(enrollment) toVisit 3 (Week 36-44) | 18.87 (18.685) | 17.10 (17.811)
  From Visit 1(enrollment) toVisit 4 (Week 56-64): number analyzed (Participants) | 794 | 270
  From Visit 1(enrollment) toVisit 4 (Week 56-64) | 20.78 (19.330) | 19.93 (20.318)

3. Primary Outcome: Change in Functional Activity of the Joint Subscale
Description: KOA patients used KOOS questionnaire, HOA patients used HOOS questionnaire. Functional activity is one subscale of KOOS and HOOS questionnaire, each functional activity question provides standard answer options: 0=None, 1=Mild, 2=Moderate, 3=Severe, 4=Extreme. The results for KOOS functional activity subscale were calculated by converting value of all subscale questions to KOOS-Physical Short form score. Results score is from 0 to 100, 100 indicating no symptoms and 0 indicating extreme symptoms. HOOS functional activity subscale results used a similar method with HOOS-Physical Short form.
Time Frame: From enrollment up to 64 weeks
Population: The outcome measure was analyzed based on participants who has KOOS/HOOS assessment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants With Stage I-III Knee Osteoarthritis (KOA) | Participants With Stage I-III Hip Osteoarthritis (HOA)
Number analyzed (Participants) | 824 | 278
Scores on a scale
  From Visit 1(enrollment) to Visit 2 (Week 16-24): number analyzed (Participants) | 798 | 272
  From Visit 1(enrollment) to Visit 2 (Week 16-24) | 10.98 (11.831) | 13.26 (15.729)
  From Visit 1(enrollment) to Visit 3 (Week 36-44): number analyzed (Participants) | 794 | 271
  From Visit 1(enrollment) to Visit 3 (Week 36-44) | 14.26 (13.708) | 16.41 (16.584)
  From Visit 1(enrollment) to Visit 4 (Week 56-64): number analyzed (Participants) | 794 | 270
  From Visit 1(enrollment) to Visit 4 (Week 56-64) | 16.60 (14.503) | 18.77 (18.041)

4. Primary Outcome: Change in Life Quality Subscale
Description: KOA patients used KOOS questionnaire, HOA patients used HOOS questionnaire. Life quality is one subscale of KOOS and HOOS questionnaire, each life quality question provides standard answer options: 0=None, 1=Mild, 2=Moderate, 3=Severe, 4=Extreme. The results for KOOS life quality subscale were calculated as [100 - (mean value of all subscale questions * 100) / 4]. Results score is from 0 to 100. 100 indicating no symptoms and 0 indicating extreme symptoms. HOOS life quality subscale results calculation used a similar method.
Time Frame: From enrollment up to 64 weeks
Population: The outcome measure was analyzed based on participants who has KOOS/HOOS assessment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants With Stage I-III Knee Osteoarthritis (KOA) | Participants With Stage I-III Hip Osteoarthritis (HOA)
Number analyzed (Participants) | 824 | 278
Scores on a scale
  From Visit 1(enrollment) to Visit 2 (Week 16-24): number analyzed (Participants) | 798 | 272
  From Visit 1(enrollment) to Visit 2 (Week 16-24) | 16.29 (17.888) | 14.25 (18.068)
  From Visit 1(enrollment) to Visit 3 (Week 36-44): number analyzed (Participants) | 794 | 271
  From Visit 1(enrollment) to Visit 3 (Week 36-44) | 20.79 (19.625) | 18.82 (18.915)
  From Visit 1(enrollment) to Visit 4 (Week 56-64): number analyzed (Participants) | 794 | 270
  From Visit 1(enrollment) to Visit 4 (Week 56-64) | 24.87 (21.055) | 22.71 (21.444)

5. Secondary Outcome: Number of Participant Compliance With Drug Utilization of Theraflex
Description: Drug utilization of Theraflex as reported by the patient to their physician. Administration duration categories are: 1.patients receiving Theraflex up to 1 month inclusive; 2.patients taking Theraflex during 1 to 3 months; 3.patients taking Theraflex during 3 to 6 months; 4. patients taking Theraflex during more than 6 months. Investigators assessed compliance with the recommendations for the duration of Theraflex.
Time Frame: From enrollment up to 64 weeks
Measure: Number; unit: Participant
Arm/Group | Participants With Stage I-III Knee Osteoarthritis (KOA) | Participants With Stage I-III Hip Osteoarthritis (HOA)
Number analyzed (Participants) | 824 | 278
Participant
  Participant followed the recommendations | 753 | 253
  Participant not followed the recommendations | 59 | 21
  No data available | 12 | 4

6. Secondary Outcome: Change in Patient Satisfaction Assessment
Description: Patient satisfaction questionnaire was filled out during the visit to a doctor. A patient assessed treatment satisfaction against the Likert response scale : 5-very satisfied, 4-Satisfied, 3- No answer, 2-Dissatisfied, 1-very dissatisfied
Time Frame: From enrollment up to 64 weeks
Population: The outcome measure was analyzed based on participants who has KOOS/HOOS assessment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants With Stage I-III Knee Osteoarthritis (KOA) | Participants With Stage I-III Hip Osteoarthritis (HOA)
Number analyzed (Participants) | 824 | 278
Scores on a scale
  From Visit 1(enrollment) to Visit 2 (Week 16-24): number analyzed (Participants) | 798 | 272
  From Visit 1(enrollment) to Visit 2 (Week 16-24) | 0.8 (0.84) | 0.8 (0.87)
  From Visit 1(enrollment) to Visit 3 (Week 36-44): number analyzed (Participants) | 794 | 271
  From Visit 1(enrollment) to Visit 3 (Week 36-44) | 0.8 (0.89) | 0.9 (0.81)
  From Visit 1(enrollment) to Visit 4 (Week 56-64): number analyzed (Participants) | 794 | 270
  From Visit 1(enrollment) to Visit 4 (Week 56-64) | 0.9 (0.94) | 0.9 (0.94)

7. Secondary Outcome: Number of Participant With Concomitant Therapy of the Target Joint Osteoarthritis (OA)
Description: Concomitant therapy of the target joint osteoarthritis (OA) by choosing any of the following categories: 'Symptomatic therapy with analgesics for the target joint OA', 'Other drug treatment for pain syndrome of the target joint OA', 'Other therapy for the target joint OA'.
Time Frame: From enrollment up to 64 weeks
Measure: Number; unit: Participant
Arm/Group | Participants With Stage I-III Knee Osteoarthritis (KOA) | Participants With Stage I-III Hip Osteoarthritis (HOA)
Number analyzed (Participants) | 824 | 278
Participant
  Symptomatic therapy with analgesics for the target joint OA | 274 | 103
  Other drug treatment for pain syndrome of the target joint OA | 84 | 25
  Other therapy for the target joint OA | 36 | 4

8. Secondary Outcome: Number of Participant With Concomitant Therapy of the Target Joint Osteoarthritis (OA) Used After the Completion of Treatment With Theraflex
Description: as for outcome 7
Time Frame: From enrollment up to 64 weeks
Measure: Number; unit: Participant
Arm/Group | Participants With Stage I-III Knee Osteoarthritis (KOA) | Participants With Stage I-III Hip Osteoarthritis (HOA)
Number analyzed (Participants) | 824 | 278
Participant
  Symptomatic therapy with analgesics for the target joint OA | 20 | 5
  Other drug treatment for pain syndrome of the target joint OA | 11 | 6
  Other therapy for the target joint OA | 9 | 0

ADVERSE EVENTS:
Time Frame: After initial administration of Theraflex up to 64 weeks.
Arm/Group | Participants With Stage I-III Hip Osteoarthritis (HOA) | Participants With Stage I-III Knee Osteoarthritis (KOA)
All-Cause Mortality (participants affected / at risk) | 0/278 | 1/824
Serious Adverse Events (participants affected / at risk) | 6/278 | 8/824
Other Adverse Events (participants affected / at risk) | 28/278 | 55/824
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Stage I-III Hip Osteoarthritis (HOA) (N=278) | Participants With Stage I-III Knee Osteoarthritis (KOA) (N=824)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Radicular pain (Nervous system disorders) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Stage I-III Hip Osteoarthritis (HOA) (N=278) | Participants With Stage I-III Knee Osteoarthritis (KOA) (N=824)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 12 (12)
Respiratory tract infection (Infections and infestations) | 7 (7) | 18 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 9 (10)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5)
Headache (Nervous system disorders) | 3 (5) | 11 (11)
Hypertension (Vascular disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-07-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT03330288/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT03330288/SAP_001.pdf